CLINICAL TRIAL: NCT06646029
Title: Pilot Study on The Effectiveness of Relative Motion Orthosis in Finger Motion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-00609
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Proximal Interphalangeal Joint Stiffness
MeSH Terms: interventions — Splints; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Orthosis + standard hand therapy care (Experimental): Patients will receive a custom splint/orthosis will be made by the hand therapist for patients to wear through the day for the length of the treatment as much as possible in additional to standard of care hand therapy. Patients will be encouraged use the orthosis during the day (at least 6-8 hours) for 6 weeks.
  Interventions: Device: RMO flexion orthosis (splint); Other: Standard of care
- Standard of care (Active Comparator): Standard of care (control group) will only complete the routine treatment. This consists of physical therapy exercises, stretches, manual therapy and use of therapeutic modalities.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: RMO flexion orthosis (splint) — RMO flexion is an orthosis fabricated by hand therapists made of thermoplastic material design to position the involved finger in relative flexion at the metacarpal joint compared to adjacent fingers to facilitate PIP extension during daily activity use.
  Arms: Orthosis + standard hand therapy care
Other: Standard of care — Treatment includes finger stretches, active range of motion (AROM), passive range of motion (PROM), thermal modalities, LMB finger extension orthosis.

SUMMARY:
The purpose of this feasibility pilot study is to determine the effectiveness of Relative Motion Orthosis (RMO) in regaining finger range of motion compared to standard care in patients diagnosed with Proximal Interphalangeal (PIP) stiffness with an extension lag secondary to finger injury. Participants will be enrolled and randomized into groups receiving either standard conservative interventions or standard interventions in addition to the RMO. The primary endpoint is to evaluate the efficacy of relative motion orthosis in PIP ROM using clinical scoring and physical exam findings.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-80
* Any gender
* Any Proximal Interphalangeal (PIP) injury that causes reduced PIP Active Range of Motion (AROM) in extension
* Right or left hand injury
* Level of Chronicity (4 weeks - 6 months)
* Able to follow instructions

Exclusion Criteria:

* PIP with hard end feel (feels they need serial casting) - level of chronicity
* Any digital nerve injury / skin laceration that can prevent the patient from using the orthosis
* Severe arthropathy
* Literacy deficits: patients need to be able to follow verbal and written instructions independently to minimize risks and improve outcomes from care.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in QuickDASH (Disability of the Arm, Shoulder, and Hand) score | Baseline, End-of-treatment (~Month 3)
  The QuickDASH Questionnaire consists of 30 items where each question in the scale is scored between 1 and 5. The total score ranges from from 0 (no difficulty or symptoms) to 100 (no activity or very severe symptoms). A decrease from baseline indicates improvement in symptoms.

SECONDARY OUTCOMES:
Change in Active Range of Motion (AROM) | Baseline, End-of-treatment (~Month 3)
  Active Range of Motion (AROM) measurement will be evaluated using a universal goniometer. The goniometer is placed at the joint, and the joint is moved through its range of motion. The goniometer measures the angle in degrees, ranging from 0 to 180. An increase from baseline indicates improved range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Ruiz, DPT, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The de-identified participant data from the final research dataset will be shared to achieve aims in the approved proposal beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Natalia.Ruiz@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.